CLINICAL TRIAL: NCT00683865
Title: Prospective, Randomized, Double-blind, Multicenter, Multinational Study Comparing Efficacy and Safety of Moxifloxacin 400 mg po od for 14 Days With Ofloxacin 400 mg po Bid Plus Metronidazole 500 mg po Bid for 14 Days in Patients With Uncomplicated Pelvic Inflammatory Disease (PID)
Brief Title: Uncomplicated Pelvic Inflammatory Disease. Treatment With Moxifloxacin.
Acronym: MAIDEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10995
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Pelvic Inflammatory Disease
Keywords: Antibiotic treatment; Pelvic infection; Interventional study; Female
MeSH Terms: conditions — Pelvic Inflammatory Disease; Pelvic Infection | interventions — Ofloxacin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Ofloxacin
- Arm 2 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)

INTERVENTIONS:
Drug: Ofloxacin — Ofloxacin 400 mg po bid plus metronidazole 500 mg po bid for 14 days
  Arms: Arm 1
Drug: Avelox (Moxifloxacin, BAY12-8039) — Moxifloxacin 400 mg po od for 14 days
  Arms: Arm 2

SUMMARY:
Comparison of various antibiotics in treatment of uncomplicated pelvic inflammatory disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PID based on: pelvic discomfort- Direct lower abdominal tenderness;
* Adnexal tenderness on bimanual vaginal examination,
* Temperature > 38.0°C; - Elevated C-reactive protein value (CRP);
* Signed PIC/IC

Exclusion Criteria:

* Pregnancy
* Abnormal lab values

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2003-04; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Clinical response 5 to 24 days after the last dose of study medication | 5 to 24 days after the last dose

SECONDARY OUTCOMES:
Bacterial response at the test of cure visit and at the FU visit 28 to 42 days after last dose of study medication | visit 28 to 42 days after last dose
Clinical response at during-treatment visit (Day 4-7) and at follow-up 28 to 42 days after last dose | (Day 4-7) and at follow-up 28 to 42 days after last dose
Reduction from baseline in pain report at the different assessment visits | Over the entire trial period (overall)
Necessity for modifying antibiotic therapy at the during-treatment visit and TOC visit and necessity for institution of an antibiotic therapy at follow-up | Over the entire trial period (overall)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (63):
- Denmark (3):
  - Hvidovre
  - Odense C
  - Roskilde
- Finland (4):
  - Hämeenlinna
  - Helsinki
  - Joensuu
  - Kotka
- France (15):
  - Antony
  - Beaumont
  - Bordeaux
  - Brive-la-Gaillarde
  - Cenon
  - Colombes
  - Créteil
  - Domont
  - Lille
  - Montauban
  - Montpellier
  - Muret
  - Nancy
  - Paris
  - Toulouse
- Germany (7):
  - München, Bavaria
  - Rostock, Mecklenburg-Vorpommern
  - Essen, North Rhine-Westphalia
  - Grevenbroich, North Rhine-Westphalia
  - Leverkusen, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Berlin, State of Berlin
- Greece (2):
  - Athens, Attica
  - Dourouti-Ioannina, Ioannina
- Hungary (4):
  - Budapest
  - Eger
  - Győr
  - Kecskemét
- Italy (3):
  - Pavia
  - Perugia
  - Trieste
- Lithuania (2):
  - Klaipėda
  - Vilnius
- Poland (7):
  - Bialystok
  - Krakow
  - Lodz
  - Lublin
  - Owock
  - Poznan
  - Warsaw
- Moscow, Russia
- South Africa (5):
  - Bloemfontein, Free State
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
- Sweden (5):
  - Gothenburg
  - Linköping
  - Lund
  - Trollhättan
  - Varberg
- United Kingdom (5):
  - Bristol, Avon
  - London, Greater London
  - Southampton, Hampshire
  - Nottingham, Nottinghamshire
  - Birmingham, West Midlands